CLINICAL TRIAL: NCT00680108
Title: A Double-Masked, Randomized, Placebo-Controlled, Rising-Dose Study of Multiple Ocular Instillations of INS365 Ophthalmic Solution in Patients With Mild to Moderate Dry Eye Disease.
Brief Title: A Study to Determine the Safety and Tolerability of Escalating Doses of INS365 Ophthalmic Solution
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-102
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — diquafosol; Ophthalmic Solutions

INTERVENTIONS:
Drug: diquafosol tetrasodium (INS365) ophthalmic solution

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of INS365 Ophthalmic Solution when applied topically as eyedrops in patients with mild to moderate dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity 20/40 in each eye
* 2 out 5 specified symptoms
* Corneal fluorescein staining score greater than or equal to 3 out of 15

Exclusion Criteria:

* Unable to stop concomitant medications
* Have had intraocular surgery in previous 90 days
* Have excluded systemic or ocular disease
* Wear contact lenses and are not willing to remove them
* Have intraocular pressure greater than 22 mg Hg

Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 1999-09; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse events
Ocular symptomatology
Visual acuity
Biomicroscopy
Ophthalmoscopy

SECONDARY OUTCOMES:
Unanesthetized Schirmer test

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Merck Sharp & Dohme LLC